CLINICAL TRIAL: NCT02886780
Title: Concentrated Exposure Treatment (cET) for Obsessive Compulsive Disorder (OCD). A Randomized Controlled Trial (RCT)
Brief Title: "Concentrated Exposure Treatment" (cET) for for Obsessive Compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/794 (REK vest)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2020-02

CONDITIONS: Obsessive Compulsive Disorder (OCD)
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Concentrated Exposure Treatment (cET) (Experimental): Please refer to:Havnen, A., Hansen, B., Öst, L.-G. & Kvale, G. Concentrated ERP delivered in a group setting: An effectiveness study. Journal of Obsessive Compulsive and Related Disorders 3, 319-324 (2014)
  Interventions: Behavioral: Concentrated exposure treatment (cET)
- Self-help (Active Comparator): The self-help condition (SH):
  Foa, E.B. & Kozak, M.J. Mastery of obsessive-compulsive disorder: Client workbook, (Graywind Publications, New York, 1997).
  Interventions: Behavioral: Self-help
- Wait list (No Intervention)

INTERVENTIONS:
Behavioral: Concentrated exposure treatment (cET) — Psychological cognitive behavioral treatment
  Arms: Concentrated Exposure Treatment (cET)
Behavioral: Self-help
  Arms: Self-help

SUMMARY:
Obsessive Compulsive Disorder (OCD) often becomes chronic if not treated. Exposure and response prevention (ERP) is recommended psychological treatment. The OCD-team at Haukeland University hospital has developed a concentrated 4-day treatment format which has been evaluated as part of standard care. Next step in the methodological development is to conduct a randomized controlled trial where the 4-day format is compared to self-help and waiting list. The study will be conducted at Solvang DPS, Sørlandet Hospital. Participants (16 in each group) are ordinary patients (>18 yrs) entitled to care in the specialist health care.

ELIGIBILITY:
Inclusion Criteria:

OCD-patients referred to the OCD-team at Sørlandet Sykehus, Solvang DPS will be included.

Inclusion criteria

* Outpatients
* ≥ 18 years of age
* Fulfilling diagnostic criteria of OCD according to the DSM-5
* Y-BOCS ≥ 16
* Fluent in Norwegian
* Signed informed consent

Exclusion Criteria:

* OCD symptoms primarily associated with hoarding
* Ongoing substance abuse/dependence
* Bipolar disorder or psychosis
* Ongoing suicidal ideation
* Mental Retardation, based on previous medical history
* If using antidepressants:

  * Not on stable dosage 4 weeks before the intervention
  * Unwilling to remain on stable dosage during the four intervention days
* Unwilling to refrain from anxiety reducing substances, such as anxiolytics (e.g. benzodiazepines) and alcohol during the two days of exposure.
* Patients living > 1.5 hour drive by car/ train from the treatment location.
* Patients with a BMI-index considered too low for participation in psychological treatment
* Patients with a full course of prior CBT for OCD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Y-BOCS from pre cET-treatment to post treatment/ waiting list/ self-help | Pre-treatment, 1 week post, minimum nine weeks after pre-treatment, minimum six months follow up
  Y-BOCS changes will for all conditions be calculated by two approaches which will be compared.
Changes i OCD diagnostic status (DSM-5) as measured by SCID | Pre-treatment, 1 week post, minimum nine weeks after pre-treatment, minimum six months follow up

SECONDARY OUTCOMES:
Well-being | Pre-treatment, 1 week post, minimum nine weeks after pre-treatment, minimum six months follow up
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) will be administered to assess mental well-being. This scale has 14 items covering different aspects of mental health related to mental well-being.
Work and social adjustment | Pre-treatment, 1 week post, minimum nine weeks after pre-treatment, minimum six months follow up
  The Work and Social Adjustment Scale (W & SAS) is a short questionnaire measuring work and social adjustment.
Generalized anxiety | Pre-treatment, 1 week post, minimum nine weeks after pre-treatment, minimum six months follow up
  Generalized Anxiety Disorder Assessment 7 (GAD-7) is a brief 7-item self-report measure for generalized anxiety symptoms. Although developed for measuring severity of generalized anxiety disorder, the GAD-7 measures severity of general anxiety symptoms common to several anxiety disorders
Depression | Pre-treatment, 1 week post, minimum nine weeks after pre-treatment, minimum six months follow up
  Patient Health Questionnaire, (PHQ-9) is a 9-item self-report questionnaire measuring level of depressive symptoms. Items are scored on a scale from 0 (not at all) to 3 (nearly every day).
Insomnia | Pre-treatment, 1 week post, minimum nine weeks after pre-treatment, six months follow up
  The Bergen Insomnia Scale (BIS) will be used to screen for sleep disturbances. The scale has six items covering different aspects of sleep disturbances the past 4 weeks
Client satisfaction | 1 week post Concentrated Exposure Treatment
  Client Satisfaction Questionnaire (CSQ-8) is an eight-item self-report form where patients report their level of satisfaction with the treatment they have undergone.

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Kvale, PhD, Principal Investigator — Haukeland UH; Gunvor Launes, MD, Study Chair — Sorlandet Hospital HF

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Launes G, Hagen K, Sunde T, Ost LG, Klovning I, Laukvik IL, Himle JA, Solem S, Hystad SW, Hansen B, Kvale G. A Randomized Controlled Trial of Concentrated ERP, Self-Help and Waiting List for Obsessive- Compulsive Disorder: The Bergen 4-Day Treatment. Front Psychol. 2019 Nov 15;10:2500. doi: 10.3389/fpsyg.2019.02500. eCollection 2019. PMID 31803089